CLINICAL TRIAL: NCT06990672
Title: Developing and Evaluating a WeChat-based Digital Therapeutic Intervention To Enhance Postoperative Fluid Adherence In Patients With Urinary Calculi: Study Protocol
Brief Title: WeChat-Based Digital Therapy to Improve Fluid Intake in Kidney Stone Patients: Study Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Shenzhen Qianhai Shekou Free Trade Zone Hospital (Unknown)
Responsible Party: Principal Investigator, ZHOU Xue, DN Candidate, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW24-754
Record Dates: First submitted 2025-05-03; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Urinary Calculi; Postoperative Care; Chronic Disease Prevention
Keywords: Fluid Adherence; Urinary Calculi; Digital Therapeutic; WeChat Applet; Post-operative
MeSH Terms: conditions — Urinary Calculi | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Receive the same standard dietary counseling and education handout but also the WeChat applet intervention. A WeChat-based applet will be developed for fluid intake adherence improvement and self-monitoring to prevent urinary calculi, including fluid intake reminders, fluid value recording, urine value and color recording, health education, an interactive platform for urinary stone prevention among post-operative patients with urinary stones. The WeChat applet will tailor the daily notification to participants of fluid intake to increase their daily fluid consumption to more than 2,500 ml. Extra education information regarding the benefits of adherence will be provided to the experimental group only via the applet. Phone calls will be given at each follow-up phase to collect primary and secondary data via the questionnaires.
Who Masked: Outcomes Assessor
Masking Description: To ensure the integrity and objectivity of outcome assessments in this randomized controlled trial, independent outcomes assessors, who are masked to participants' group assignments, will be employed. These assessors, comprising trained research nurses and clinical research coordinators not involved in the delivery of the WeChat applet intervention or usual care, will be responsible for evaluating primary and secondary outcomes. Masking will be maintained through secure data management systems that conceal group allocation (WeChat applet vs. usual care) during data collection and analysis. The assessors will receive training on standardized outcome measurement protocols and will have no direct interaction with participants or intervention staff to prevent unmasking. This approach minimizes assessment bias, enhancing the reliability of trial results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Other): Standard care or usual care such as receiving standard dietary and verbal education counselling will be delivered in this arm
  Interventions: Other: Standard care
- WeChat Applet Intervention (Experimental): WeChat Applet intervention involving both standard care and WeChat applet will be delivered to the experimental arm
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Standard care — Receiving standard dietary and regular recommendations such as education profile and counseling to achieve a fluid intake ≥ 2500 ml, providing verbal health education counseling regarding urological calculi prevention during the hospitalization, and adequate fluid intake in person on the day of discharge. Prepare a fixed-capacity water bottle. Phone calls will be given at each follow-up phase to collect primary and secondary data via the questionnaires.
  Arms: Standard care
Other: Experimental — Receive the same standard dietary counseling and education handout but also the WeChat applet intervention. A WeChat-based applet will be developed for fluid intake adherence improvement and self-monitoring to prevent urinary calculi, including fluid intake reminders, fluid value recording, urine value and coluor recording, and health education, an interactive platform for communication among post-operative patients with urinary stones. The applet will tailor the daily notification to participants of fluid intake to increase their fluid consumption to more than 2,500 ml. Extra education information regarding the benefits of adherence will be provided to the experimental group only via the applet. Phone calls will be given at each follow-up phase to collect primary and secondary data via the questionnaires.
  Arms: WeChat Applet Intervention

SUMMARY:
The goal of this clinical trial is to learn Whether the WeChat-based applet works to prevent urinary calculi for postoperative patients. The main questions it aims to answer are:

Dose the WeChat-based applet intervention increase the amount of fluid intake and urine output? Researchers will compare the WeChat-based applet intervention to a usual care to see if the WeChat-based applet works to prevent urinary calculi occurence.

Participants will:

1. Using the WeChat-based applet or a placebo every day for 3 months
2. Keep a record of their fluid intake, urine output, number of urinary calculi recurrence

DETAILED DESCRIPTION:
The study outcomes will be reported to adhere to the guidelines outlined in the Consolidated Standards of Reporting Trials (CONSORT) 2010 statements. Reporting measures of central tendency (mean, median) and dispersion (standard deviation, range) for continuous variables, as well as frequencies and percentages for categorical variables. Statistical tests such as a t-test and chi-square test will be employed for continuous and categorical variables within two groups. The principal analysis will compare the fluid intake volume between the intervention and control groups using the t-test. Secondary outcomes such as The Wisconsin Stone Quality of Life Questionnaire (WISQOL), Patient Health Questionnaire-9 Items (PHQ-9), International Physical Activity Questionnaire (IPAQ-SF ) and The Electronic Health Literacy Scale (eHEALS) will use repeated measures of Analysis of Variance (ANOVA) since they are measured over time and between two groups. If necessary, subgroup analyses will be conducted to explore whether the effect of the intervention varies across different demographic or clinical subgroups. Intention-to-treat (ITT) analysis will be used to assess the impact of the treatment and its generalizability. A significance level of p < 0.05 will be utilized to determine statistical significance, and all data analysis procedures will be conducted using the SPSS (Statistical Product and Service Solutions) 26.0 software package.The researcher is granted access to the complete trial dataset, with a contractual agreement established with the statistician to manage the data confidentially in accordance with the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* With a history of urinary calculi and having received urolithiasis surgery before
* 24-hour fluid intake < 2500 ml
* Age ≥ 18 years old
* Able to use WeChat daily
* Able to read and write informed consent

Exclusion Criteria:

* Participants with obstructive uropathy, chronic urosepsis, renal failure, and renal tubular acidosis
* Participants with congestive heart failure, psychiatric conditions, pregnancy, and primary hyperparathyroidism
* Participants experienced complicated urolithiasis surgery.
* History of recurrent UTI (urinary tract infection) (>3/year)
* Medication use increases stone risk.
* Participants with physical disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and Male
Enrollment: 148 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
24-hour urine volume (ml) | Up to three months
  24-hour urine volume (ml) ： Measurement method: Participants will void into a calibrated container upon waking in the morning and record the precise start time (e.g., 8:00 AM). At the same time point 24 hours later, urine volume will be remeasured. Cumulative urine output will be tracked using a WeChat-based applet or alternative recording tools.
24-hour fluid intake volume (ml) | Up to three months
  24-hour fluid intake volume (ml) ： Measurement method: Participants will record all fluid consumption (including water, tea, coffee, herbal tea, and other eligible liquids) over a standardized 24-hour period using a WeChat-based applet. Recording will begin and end at the same time daily.

SECONDARY OUTCOMES:
Wisconsin Stone Quality of Life Questionnaire (WISQOL) | Up to three months
  Scale range: A 5-point scale from 1 to 5 yielding a total score range between 28 and 140 points, a higher score indicates a better quality of life
Patient Health Questionnaire-9 items (PHQ-9) | Up to three months
  9 items with a cumulative score on the PHQ-9 range from 0 to 27 points, the higher score represented a greater severity of depressive symptoms;
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | [Time Frame: Up to three months]
  score Calculation: Metabolic Equivalent of Task (MET) = MET value (3.3-8) × activity duration (minutes) × frequency (days) Classification: <600 MET-min/week = low activity; 600-3000 MET-min/week = middle activity; >3000 MET-min/week = high activity
eHealth Literacy Scale (eHEALS) | Up to three months
  A scale including 8 items with a five-point Likert scale; Scale range: 8-40 points (higher scores indicate better eHealth literacy)
Number of outpatient visits or readmission | Up to three months
  The number of outpatient visits is defined as the frequency of medical consultations during the study period due to urinary calculi-related symptoms (e.g., hematuria, pain) or complications (e.g., urinary tract infections). Readmission is defined as hospitalization events resulting from stone recurrence, severe complications, or surgical requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Datas collect from Primary outcome such as 24-hour urine volume (ml);24-hour fluid intake volume (ml) and secondary outcome such as The Wisconsin Stone Quality of Life Questionnaire (WISQOL);PHQ-9 (patient health questionnaire-9 items);IPAQ-SF (International Physical Activity Questionnaire);The eHEALS (Electronic Health Literacy Scale);The number of outpatient visits; recurrence rate will be shared. Part of the demographic data such as the time of using WeChat, gender, age, the type of surgery and BMI will shared.
Supporting Information: ICF
Time Frame: The data will be available for 3 years:
  The start date: 1 Dec 2025; The end date: 30 Nov 2028.
Access Criteria: IPD and supporting information collected in this study will be accessible exclusively to accredited researchers. These researchers must be members of academic institutions or research organizations relevant to the field of this study and possess a clear research purpose along with a rational analysis plan. Additionally, researchers are required to sign a data use agreement to ensure the confidentiality and compliant use of the data.
  Content Available for Access:
  Researchers will have access to de-identified IPD, encompassing participants' baseline characteristics, interventions, follow-up data, and primary and secondary outcome measures. Supporting information, such as the study protocol and statistical analysis plan, will also be provided to aid researchers in understanding the data structure and analysis methods.
  Mechanism of Access:
  Data access will be facilitated through a secure online data-sharing platform. Researchers are required to register and submit data access application.

REFERENCES:
- [Background] 1. Shafi, H., et al., An overview of treatment options for urinary stones. Caspian journal of internal medicine, 2016. 7(1): p. 1. 2. Sorokin, I., et al., Epidemiology of stone disease across the world. World journal of urology, 2017. 35: p. 1301-1320. 3. Romero, V., H. Akpinar, and D.G. Assimos, Kidney stones: a global picture of prevalence, incidence, and associated risk factors. Reviews in urology, 2010. 12(2-3): p. e86. 4. Zeng, G., et al., Prevalence of kidney stones in China: an ultrasonography based cross-sectional study. BJU international, 2017. 120(1): p. 109-116. 5. Johnson, C.M., et al., Renal stone epidemiology: a 25-year study in Rochester, Minnesota. Kidney international, 1979. 16(5): p. 624-631. 6. Pearle, M.S., et al., Urologic diseases in America project: urolithiasis. The Journal of urology, 2005. 173(3): p. 848-857. 7. Moftakhar, L., et al., Prevalence and risk factors of kidney stone disease in population aged 40-70 years old in Kharameh cohort study: a cross-sectional population-based study in southern Iran. BMC urology, 2022. 22(1): p. 205. 8. Fakheri, R.J. and D.S. Goldfarb, Ambient temperature as a contributor to kidney stone formation: implications of global warming. Kidney international, 2011. 79(11): p. 1178-1185. 9. Becerra, A.Z., et al., Contemporary assessment of the economic burden of upper urinary tract stone disease in the United States: analysis of one-year health care costs, 2011-2018. Journal of Endourology, 2022. 36(4): p. 429-438. 10. Lotan, Y., et al., Primary prevention of nephrolithiasis is cost-effective for a national healthcare system. BJU international, 2012. 110(11c): p. E1060-E1067. 11. Mitra, P., D.K. Pal, and M. Das, Does quality of drinking water matter in kidney stone disease: A study in West Bengal, India. Investig Clin Urol, 2018. 59(3): p. 158-165. 12. Mathiyalagen, P., et al., A case-control study on environmental and biological risk factors for renal calculi persisting in a coastal Union Territory, India.